CLINICAL TRIAL: NCT01467674
Title: Malondialdehyde And Antioxidant Levels In Chronic Periodontitis Patients With Type 2 Diabetes Mellitus Under Different Stages Of Metabolic Control
Brief Title: The Effect Of Glycemic Control On Malondialdehyde, Glutathione Peroxidase, Glutathione And Paraoxonase
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Dr. Yener ÖZAT, Assistant Professor, Suleyman Demirel University
Other Study IDs: 1721-D-08
Record Dates: First submitted 2011-11-01; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Periodontitis
Keywords: Diabetes mellitus; Chronic periodontitis; Malondialdehyde; Glutathione peroxidase; Paraoxonase
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy
- Chronic Periodontitis
- Better Controlled T2DM
- Poor Controlled T2DM

SUMMARY:
The aim of this study was to investigate the impact of glycemic control on clinical periodontal status, levels of malondialdehyde (MDA), glutathione peroxidase (GSH-Px), reduced glutathione (GSH) and paraoxonase (PON) activity in gingival crevicular fluid (GCF) and blood samples of type 2 diabetes mellitus (T2DM) patients with chronic periodontitis (CP).

DETAILED DESCRIPTION:
Reactive oxygen species (ROS) are products of normal cellular metabolism and play beneficial role in physiological functions. Overproduction of ROS and/or deficiency of enzymatic or non-enzymatic antioxidants, termed as oxidative stress, is involved in many pathological conditions such as Diabetes mellitus (DM) and chronic periodontitis (CP).

Several researches revealed that DM, with many determinants such as level of glycemic control, stands as a strong risk factor for periodontal diseases. On the other side, periodontal diseases induce an elevated chronic inflammatory state and exacerbated insulin resistance.

In the present study, the investigators examined the effect of glycemic control level on clinical periodontal status, levels of MDA, GSH-Px, GSH and PON activity in gingival crevicular fluid and blood samples of CP patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* to present T2DM diagnosis by an endocrinologist for at least the past 5 years
* diagnosis of CP was based on the clinical and radiographic criteria proposed by the 1999 World Workshop for Classification of Periodontal Diseases and Conditions

Exclusion Criteria:

* pregnancy
* lactation
* current smoking or smoking within the past 2 years, periodontal therapy in the previous 6 months
* antibiotic and/or antimicrobial therapies in the previous 3 months
* existence of serious diabetic complications or any pathology such as haemoglobinopathy which would affect haemoglobin profile
* diagnosis of another major medical pathology, middle or upper-level obesity according to WHO classification
* current anti-hyperlipidemic therapy
* non-T2DM patients with abnormal values of glucose and lipid metabolism parameters, major medical pathology and family history of DM

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with T2DM were recruited among those attending Suleyman Demirel University (SDU) Faculty of Medicine, Department of Endocrinology and non-diabetic individuals were recruited among those attending SDU Faculty of Dentistry, Department of Periodontology.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | One Year
  Level of Metabolic Control

SECONDARY OUTCOMES:
Clinical Periodontal Status | One Year
  Periodontal indices evaluating clinical periodontal health status

CONTACTS AND LOCATIONS:
Overall Officials: F. Yeşim Kırzıoğlu, 1, Study Director — Professor, Periodontology Dept; Mustafa Nazıroğlu, 1, Study Director — Professor, Biophysics Dept; M. Numan Tamer, 1, Study Director — Professor, Internal Diseases Dept.
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)